CLINICAL TRIAL: NCT05541718
Title: New Options for Treating Knee Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00153103
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutic Touch; Mindfulness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reiki (Experimental)
  Interventions: Behavioral: Reiki
- Sham Reiki (Sham Comparator)
  Interventions: Behavioral: Sham Reiki
- Mindfulness Meditation (Active Comparator)
  Interventions: Behavioral: Mindfulness Meditation
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Reiki — Reiki will be provided by a trained Reiki master with the aim of balancing the flow of energy in the patient's body.
  Arms: Reiki
Behavioral: Sham Reiki — Sham Reiki will be delivered by an individual trained to simulate the Reiki interventionist's movements, but they will not visualize patient healing
  Arms: Sham Reiki
Behavioral: Mindfulness Meditation — The mindfulness meditation intervention will be adapted from a standardized mindfulness induction script validated in prior research. The mindfulness practice will guide patients to focus attention on breath and body sensations while monitoring and accepting discursive thoughts, negative emotions, and pain. The MM interventionist will be a trained mindfulness provider and have experience using MM in medical settings.
  Arms: Mindfulness Meditation

SUMMARY:
This study will be a single-site, four-arm, randomized, placebo-controlled clinical trial. Knee osteoarthritis patients (N=164) will be randomized to Reiki, Sham Reiki (placebo control), mindfulness meditation (active control), or a waitlist control condition. The three active interventions will be applied for 20 minutes, once a week, for four consecutive weeks in a university laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis in at least one knee
* Report a WOMAC pain score average >/= 2
* Not using any kind of energy therapy different from the proposed study
* Ability to read, understand and speak English

Exclusion Criteria:

* Knee arthroplasty in the previous year
* Have cognitive impairment as determined by clinical interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Change in Osteoarthritis symptoms | One week before treatment to one week after treatment, which comprises a 6 week span
  The Western Ontario and McMaster Universities Arthritis Index will be used to measure change in osteoarthritis symptoms. Scores range from 0 to 96, with higher scores reflect worse pain, stiffness and physical function

SECONDARY OUTCOMES:
Change in Depression | One week before treatment to one week after treatment, which comprises a 6 week span
  The Patient Health Questionnaire-2 will be used to measure depression. Scores range from 0 to 6, with higher scores reflect worse depression
Change in Anxiety | One week before treatment to one week after treatment, which comprises a 6 week span
  The Generalized Anxiety Disorder 2-item will be used to measure anxiety. Scores range from 0 to 6, with higher scores reflect worse anxiety.
Change in Pain Catastrophizing | One week before treatment to one week after treatment, which comprises a 6 week span
  The Pain Catastrophizing Scale will be used to measure pain catastrophizing. Scores range from 0 to 52, with higher scores reflect worse pain catastrophizing
Change in Sleep | One week before treatment to one week after treatment, which comprises a 6 week span
  The PROMIS Sleep Disturbance - Short Form 6a will measure changes in sleep. Scores range from 0 to 30, with higher scores reflect greater sleep disturbance
Change in Quality of Life | One week before treatment to one week after treatment, which comprises a 6 week span
  The WHOQOL-BREF will measure quality of life. Scores range from 0 to 100, with higher scores reflect better quality of life
Change in Acute Pain Intensity | Immediately before to after the first and last treatment session, which comprises a 20 minute span
  Single item assessing pain intensity ("How much pain do you have?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain intensity.

OTHER OUTCOMES:
Change in State Self-Transcendence | Immediately before to after the first and last treatment session, which comprises a 20 minute span
  Change in self-transcendent state will be measured with the Nondual Awareness Dimensional Assessment - State Version. Scores range from 0 to 10, with higher scores reflecting greater self-transcendence.
Change in State Decentering | Immediately before to after the first and last treatment session, which comprises a 20 minute span
  Change in state decentering will be measured with the Metacognitive Processes of Decentering Scale - State Version. Scores range from 0 to 10, with higher scores reflecting greater state decentering.
Change in Trait Self-Transcendence | One week before treatment to one week after treatment, which comprises a 6 week span
  Change in trait self-transcendence will be assessed with the Nondual Awareness Dimensional Assessment - Trait Version. Scores range from 0 to 10, with higher scores reflecting greater trait self-transcendence.
Change in Trait Decentering | One week before treatment to one week after treatment, which comprises a 6 week span
  Change in trait decentering will be assessed with the Metacognitive Processes of Decentering Scale - Trait Version. Scores range from 0 to 10, with higher scores reflecting greater trait decentering.
Change in Prescription Pain Medication Misuse | One week before treatment to one week after treatment, which comprises a 6 week span
  The PROMIS Prescription Pain Medication Misuse v1.0 - Short Form 7a will measure prescription pain medicine misuse. Scores range from 0 to 35, with higher scores reflecting greater misuse.
Pleasant Sensation Ratio | Immediately before to after the first and last treatment session, which comprises a 20 minute span
  Pleasant sensation ratio as measured by Sensation Manikin, a measure comprised of a visual body map to demonstrate the location and distribution of sensations.
Quantitative sensory testing | Immediately before the first treatment session and immediately after the last treatment session, which comprises a 4 week span
  Pain threshold and tolerance, temporal summation, and conditioned pain modulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05541718/SAP_001.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05541718/ICF_000.pdf